CLINICAL TRIAL: NCT02643342
Title: A 2-year Longitudinal Study on the Structural and Optical Effects of Orthokeratology Treatment on Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry); Queensland University of Technology (Other); Aston University (Other)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20150909002
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-02

CONDITIONS: Myopic Progression
Keywords: myopia control; orthokeratology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single-vision glasses (No Intervention): Subjects wearing single-vision glasses CR-39 of refractive index 1.56.
- Orthokeratology with normal compression factor (Sham Comparator): Subjects wearing orthokeratology lenses of normal compression factor about 0.50-0.75D.
  Interventions: Device: Orthokeratology
- Orthokeratology with increased compression factor (Active Comparator): Subjects wearing orthokeratology lenses of increased compression factor about 1.50-1.75D.
  Interventions: Device: Orthokeratology

INTERVENTIONS:
Device: Orthokeratology
  Other Names: ortho-k
  Arms: Orthokeratology with increased compression factor; Orthokeratology with normal compression factor

SUMMARY:
This is a two-year longitudinal study investigating the optical and structural effects of increased compression factor of orthokeratology lens on eyes and the corresponding effect on change in choroidal thickness and therefore myopic control.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 10 years old
* Myopia: between 0.50 D and 4.00 D in both eyes
* Astigmatism: <1.50 D; ≤ 1.25 D for with-the-rule astigmatism (axes 180 ± 30); ≤ 0.50 D for astigmatism of other axes in both eyes
* Anisometropia: ≤ 1.50 D
* Symmetrical corneal topography with corneal toricity <2.00 D in both eyes
* Agree for randomization

Exclusion Criteria:

* Contraindications for orthokeratology wear (e.g. limbus-to-limbus corneal cylinder and dislocated corneal apex)
* Any type of strabismus or amblyopia
* Myopic treatment (e.g. refractive surgery and progressive lens wear for myopic control) before and during the study period
* Rigid contact lenses (including orthokeratology lenses) experience
* Systemic condition which might affect refractive development (for example, Down syndrome, Marfan's syndrome)
* Ocular conditions which might affect the refractive error (for example, cataract, ptosis)
* Poor compliance for lens wear or follow-up

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2016-06-18 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2019-08-03 (Actual)

PRIMARY OUTCOMES:
Axial length | every 6 monthly in 2 years
  axial progression of the eyeball

SECONDARY OUTCOMES:
Ocular aberration measured by Complete Ophthalmic Analysis System (COAS) aberrometer | every 6 monthly in 2 years
  ocular aberration measured by Complete Ophthalmic Analysis System (COAS) aberrometer
Corneal biomechanics (corneal response using ocular response) | every 6 monthly in 2 years
  corneal response using ocular response
Accommodation lag measured by Complete Ophthalmic Analysis System (COAS) aberrometer | every 6 monthly in 2 years
  accommodation lag measured by Complete Ophthalmic Analysis System (COAS) aberrometer using different accommodation targets
Choroidal thickness captured by Optical Coherent Tomographer (OCT) | every 6 monthly in 2 years
  choroidal thickness captured by Optical Coherent Tomographer (OCT) and measured using a customized software

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong KOng Polytechnic University, Hong Kong, China

REFERENCES:
- [Background] Lam CS, Lam CH, Cheng SC, Chan LY. Prevalence of myopia among Hong Kong Chinese schoolchildren: changes over two decades. Ophthalmic Physiol Opt. 2012 Jan;32(1):17-24. doi: 10.1111/j.1475-1313.2011.00886.x. PMID 22150587
- [Background] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Background] Cho P, Cheung SW. Retardation of myopia in Orthokeratology (ROMIO) study: a 2-year randomized clinical trial. Invest Ophthalmol Vis Sci. 2012 Oct 11;53(11):7077-85. doi: 10.1167/iovs.12-10565. PMID 22969068
- [Background] Chen C, Cheung SW, Cho P. Myopia control using toric orthokeratology (TO-SEE study). Invest Ophthalmol Vis Sci. 2013 Oct 3;54(10):6510-7. doi: 10.1167/iovs.13-12527. PMID 24003088
- [Background] Gonzalez-Meijome JM, Villa-Collar C, Queiros A, Jorge J, Parafita MA. Pilot study on the influence of corneal biomechanical properties over the short term in response to corneal refractive therapy for myopia. Cornea. 2008 May;27(4):421-6. doi: 10.1097/ICO.0b013e318164e49d. PMID 18434845
- [Background] Wolffsohn JS, Safeen S, Shah S, Laiquzzaman M. Changes of corneal biomechanics with keratoconus. Cornea. 2012 Aug;31(8):849-54. doi: 10.1097/ICO.0b013e318243e42d. PMID 22495031
- [Background] Tse DY, Lam CS, Guggenheim JA, Lam C, Li KK, Liu Q, To CH. Simultaneous defocus integration during refractive development. Invest Ophthalmol Vis Sci. 2007 Dec;48(12):5352-9. doi: 10.1167/iovs.07-0383. PMID 18055781
- [Background] Chan B, Cho P, Mountford J. The validity of the Jessen formula in overnight orthokeratology: a retrospective study. Ophthalmic Physiol Opt. 2008 May;28(3):265-8. doi: 10.1111/j.1475-1313.2008.00545.x. PMID 18426426
- [Derived] Wan K, Lau JK, Cheung SW, Cho P. Orthokeratology with increased compression factor (OKIC): study design and preliminary results. BMJ Open Ophthalmol. 2020 May 4;5(1):e000345. doi: 10.1136/bmjophth-2019-000345. eCollection 2020. PMID 32420450